CLINICAL TRIAL: NCT06474611
Title: Evaluation of a Patient 'nudge' on Engagement in Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Debra Ritzwoller, Senior Investigator - Economics and Cancer Research, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IMP_LungCancerScreen
Record Dates: First submitted 2024-06-20; First posted 2024-06-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Masking Description: No masking involved. This is a quality improvement project where patients who have an upcoming Primary Care visit receive an electronic or paper letter notification that they qualify for lung cancer screening and that they should talk to their dr at the upcoming visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Birth year = odd (No Intervention): No intervention, care as usual
- Birth year = even AND active on KP.org (Experimental): Has an upcoming primary care visit, qualifies for lung cancer screening based on USPSTF criteria, receives an electronic letter via KP.org informing that they qualify for LCS and reminding to talk to PCP about LCS at next visit.
  Interventions: Behavioral: Patient nudge
- Birth year = even AND not active on KP.org (Experimental): Has an upcoming primary care visit, qualifies for LCS based on USPSTF criteria, receives a mailed letter informing that they qualify for LCS and reminding to talk to provider about LCS at next visit.
  Interventions: Behavioral: Patient nudge

INTERVENTIONS:
Behavioral: Patient nudge — Patient receives an electronic or paper letter 'nudge' to talk to dr about LCS.
  Arms: Birth year = even AND active on KP.org; Birth year = even AND not active on KP.org

SUMMARY:
The purpose of this quality improvement project is to conduct and evaluate the effect of sending an electronic reminder message to patients who qualify for lung cancer screening, haven't had a screening previously, and who have an upcoming scheduled appointment with their doctor.

DETAILED DESCRIPTION:
United States Preventive Services Task Force (USPSTF) lung cancer screening (LCS) guidelines recommend LCS for those aged 50-80 with at least 20 pack-years smoking history, who currently smoke or quit within the last 15 years. In 2023, our study team found that there are approximately 6,000 - 8,000 Kaiser Permanente Colorado (KPCO) members who are unscreened and eligible for lung cancer screening (LCS). In support of KP's Population Health priority initiative to expand lung cancer screening participation for those who are eligible, our study team was selected to move this work forward in 2024 with feasible implementation opportunities for the KPCO LCS Operational/Institute for Health Research partnership at its core. The primary objective of this project is to conduct and evaluate a randomized quality improvement pragmatic intervention of a 2-arm electronic message outreach to unscreened LCS members who are eligible for LCS and who have an upcoming scheduled Primary Care Provider (PCP) visit.

ELIGIBILITY:
Inclusion Criteria: Qualifies for Lung Cancer Screening based on USPSTF criteria (aged 50-80, at least 20 pack years smoking history, currently smoke or quit in the last 15 years); have an upcoming, scheduled Primary Care visit in a KP clinic in the coming 7-14 days, have not completed a low-dose CT scan.

Exclusion Criteria:

* None

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 894 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The proportion completed a visit with a Primary Care provider by receipt of an electronic letter or paper letter | 12 months
  The proportion completed a visit with a Primary Care provider by receipt of an electronic letter or paper letter
The proportion receiving an order to get a low-dose computed tomography (LDCT) lung cancer screen (LCS) scan by receipt of an electronic letter or paper letter | 12 months
  The proportion receiving an order to get a low-dose computed tomography (LDCT) lung cancer screen (LCS) scan by receipt of an electronic letter or paper letter
The proportion completing a low-dose computed tomography (LDCT) lung cancer screen (LCS) scan by receipt of an electronic letter or paper letter | 12 months
  The proportion completing a low-dose computed tomography (LDCT) lung cancer screen (LCS) scan by receipt of an electronic letter or paper letter

CONTACTS AND LOCATIONS:
Overall Officials: Debra Ritzwoller, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Quality Improvement study. No individual participant data will be available to other researchers.